| Low-Level Laser Therapy in the Management of Painful Hypersensitivity Caused by Molar-Incisor Hypomineralization in Children: A Triple-Blind, Placebo-Controlled Randomized Clinical Trial. |
|---|
| Identification number: NCT06426108 |

statistical analysis plan

After obtaining the results, the data will be subjected to normality analysis (Shapiro-Wilk Test) and homoscedasticity analysis (Levene's Test), which will indicate normality and homogeneity of the sample. Parametric statistical analysis will therefore be used. For all variables, a Two-Way ANOVA test and Duncan's post-hoc test will be employed to analyze comparisons between groups. The analyses will be conducted using the statistical software SPSS 20.0 (SPSS Inc., Chicago, IL, USA). All tests will be performed with a 95% confidence level ( $\alpha$  = 0.05).